CLINICAL TRIAL: NCT02897804
Title: Engineering an Online STI Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Linda Collins, Director of The Methodology Center and Distinguished Professor, Penn State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01AA022931 (NIH)
Record Dates: First submitted 2016-08-22; First posted 2016-09-13 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Sexual Behavior; Alcohol Consumption; Sexually Transmitted Diseases
Keywords: multiphase optimization strategy; college students
MeSH Terms: conditions — Sexual Behavior; Alcohol Drinking; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (32):
- Knowledge alone (Experimental): Participants will have access to the knowledge module for a period up to 3 weeks.
  Interventions: Behavioral: Knowledge alone
- Self-efficacy alone (Experimental): Participants will have access to the knowledge module plus the self-efficacy module for a period up to 3 weeks.
  Interventions: Behavioral: Self-efficacy alone
- Perceived benefits alone (Experimental): Participants will have access to the knowledge module plus the perceived benefits module for a period up to 3 weeks.
  Interventions: Behavioral: Perceived benefits alone
- Benefits and self-efficacy (Experimental): Participants will have access to the knowledge module plus the perceived benefits and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Perceived benefits and self-efficacy
- Injunctive norms alone (Experimental): Participants will have access to the knowledge module plus the injunctive norms module for a period up to 3 weeks.
  Interventions: Behavioral: Injunctive norms
- Injunctive norms and self-efficacy (Experimental): Participants will have access to the knowledge module plus the injunctive norms and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Injunctive norms and self-efficacy
- Injunctive norms and perceived benefits (Experimental): Participants will have access to the knowledge module plus the injunctive norms and perceived benefits modules for a period up to 3 weeks.
  Interventions: Behavioral: Injunctive norms and perceived benefits
- Injunctive norms, perceived benefits,self-efficacy (Experimental): Participants will have access to the knowledge module plus the injunctive norms, perceived benefits, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Injunctive norms, perceived benefits, and self-efficacy
- Descriptive norms alone (Experimental): Participants will have access to the knowledge module plus the descriptive norms module for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive norms alone
- Descriptive norms and self-efficacy (Experimental): Participants will have access to the knowledge module plus the descriptive norms and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive norms and self-efficacy
- Descriptive norms and perceived benefits (Experimental): Participants will have access to the knowledge module plus the descriptive norms and perceived benefits modules for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive norms and perceived benefits
- Descriptive norms,perceived benefits,self-efficacy (Experimental): Participants will have access to the knowledge module plus the descriptive norms module for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive norms,perceived benefits,self-efficacy
- Descriptive norms and injunctive norms (Experimental): Participants will have access to the knowledge module plus the descriptive norms and injunctive norms modules for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive and injunctive norms
- Descriptive norms, injunctive norms,self-efficacy (Experimental): Participants will have access to the knowledge module plus the descriptive norms, injunctive norms, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive norms, injunctive norms,self-efficacy
- Descriptive and injunctive norms, benefits (Experimental): Participants will have access to the knowledge module plus the descriptive norms, injunctive norms, and perceived benefits modules for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive and injunctive norms, benefits
- Descriptive and injunctive norms, benefits,efficacy (Experimental): Participants will have access to the knowledge module plus the descriptive norms, injunctive norms, perceived benefits, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Descriptive and injunctive norms, benefits,efficacy
- Expectancies alone (Experimental): Participants will have access to the knowledge module plus the expectancies module for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies alone
- Expectancies and self-efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies and self-efficacy
- Expectancies and perceived benefits (Experimental): Participants will have access to the knowledge module plus the expectancies and perceived benefits modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies and Perceived Benefits
- Expectancies, perceived benefits, self-efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies, perceived benefits, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, perceived benefits, self-efficacy
- Expectancies and injunctive norms (Experimental): Participants will have access to the knowledge module plus the expectancies and injunctive norms modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies and injunctive norms
- Expectancies, injunctive norms, and self-efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies, injunctive norms, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, injunctive norms, and self-efficacy
- Expectancies, injunctive norms, and benefits (Experimental): Participants will have access to the knowledge module plus the expectancies, injunctive norms, and perceived benefits modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, injunctive norms, benefits
- Expectancies, injunctive norms, benefits, efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies, injunctive norms, perceived benefits, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, injunctive norms, benefits, efficacy
- Expectancies and descriptive norms (Experimental): Participants will have access to the knowledge module plus the expectancies and descriptive norms modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies and descriptive norms
- Expectancies, descriptive norms, and self-efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies, descriptive norms, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, descriptive norms, and self-efficacy
- Expectancies, descriptive norms, and benefits (Experimental): Participants will have access to the knowledge module plus the expectancies, descriptive norms, and perceived benefits modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, descriptive norms, and benefits
- Expectancies,descriptive norms, benefits, efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies, descriptive norms, perceived benefits, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies,descriptive norms, benefits, efficacy
- Expectancies, descriptive and injunctive norms (Experimental): Participants will have access to the knowledge module plus the expectancies, descriptive norms, and injunctive norms modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, descriptive and injunctive norms
- Expectancies, descr& injun norms, efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies, descriptive norms, injunctive norms, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, descr& injun norms, efficacy
- Expectancies, desc & injun norms, benefits (Experimental): Participants will have access to the knowledge module plus the expectancies, descriptive norms, injunctive norms, and perceived benefits modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies, desc & injun norms, benefits
- Expectancies,desc & injun norms,benefits,efficacy (Experimental): Participants will have access to the knowledge module plus the expectancies, descriptive norms, injunctive norms, perceived benefits, and self-efficacy modules for a period up to 3 weeks.
  Interventions: Behavioral: Expectancies,desc & injun norms,benefits,efficacy

INTERVENTIONS:
Behavioral: Knowledge alone — Increase knowledge related STIs, STI risk, alcohol impairment, condom use skills, alcohol use behavior tracking skills, testing & treatment services.
  Arms: Knowledge alone
Behavioral: Self-efficacy alone — Increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Self-efficacy alone
Behavioral: Perceived benefits alone — Increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol.
  Arms: Perceived benefits alone
Behavioral: Perceived benefits and self-efficacy — Increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Benefits and self-efficacy
Behavioral: Injunctive norms — Correct misperceptions regarding approval of alcohol misuse & sexual risk taking.
  Arms: Injunctive norms alone
Behavioral: Injunctive norms and self-efficacy — Correct misperceptions regarding approval of alcohol misuse & sexual risk taking and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Injunctive norms and self-efficacy
Behavioral: Injunctive norms and perceived benefits — Correct misperceptions regarding approval of alcohol misuse & sexual risk taking and increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Injunctive norms and perceived benefits
Behavioral: Injunctive norms, perceived benefits, and self-efficacy — Correct misperceptions regarding approval of alcohol misuse & sexual risk taking; increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Injunctive norms, perceived benefits,self-efficacy
Behavioral: Descriptive norms alone — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors.
  Arms: Descriptive norms alone
Behavioral: Descriptive norms and self-efficacy — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Descriptive norms and self-efficacy
Behavioral: Descriptive norms and perceived benefits — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors and increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol.
  Arms: Descriptive norms and perceived benefits
Behavioral: Descriptive norms,perceived benefits,self-efficacy — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Descriptive norms,perceived benefits,self-efficacy
Behavioral: Descriptive and injunctive norms — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors and correct misperceptions regarding approval of alcohol misuse & sexual risk taking.
  Arms: Descriptive norms and injunctive norms
Behavioral: Descriptive norms, injunctive norms,self-efficacy — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Descriptive norms, injunctive norms,self-efficacy
Behavioral: Descriptive and injunctive norms, benefits — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; and increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol.
  Arms: Descriptive and injunctive norms, benefits
Behavioral: Descriptive and injunctive norms, benefits,efficacy — Correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol; and Increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Descriptive and injunctive norms, benefits,efficacy
Behavioral: Expectancies alone — Decrease the expectation that alcohol is needed to have good sexual encounter.
  Arms: Expectancies alone
Behavioral: Expectancies and self-efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies and self-efficacy
Behavioral: Expectancies and Perceived Benefits — Decrease the expectation that alcohol is needed to have good sexual encounter and increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol.
  Arms: Expectancies and perceived benefits
Behavioral: Expectancies, perceived benefits, self-efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter; increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies, perceived benefits, self-efficacy
Behavioral: Expectancies and injunctive norms — Decrease the expectation that alcohol is needed to have good sexual encounter and correct misperceptions regarding approval of alcohol misuse & sexual risk taking.
  Arms: Expectancies and injunctive norms
Behavioral: Expectancies, injunctive norms, and self-efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies, injunctive norms, and self-efficacy
Behavioral: Expectancies, injunctive norms, benefits — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; and increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol.
  Arms: Expectancies, injunctive norms, and benefits
Behavioral: Expectancies, injunctive norms, benefits, efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies, injunctive norms, benefits, efficacy
Behavioral: Expectancies and descriptive norms — Decrease the expectation that alcohol is needed to have good sexual encounter and correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors.
  Arms: Expectancies and descriptive norms
Behavioral: Expectancies, descriptive norms, and self-efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies, descriptive norms, and self-efficacy
Behavioral: Expectancies, descriptive norms, and benefits — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; and increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol.
  Arms: Expectancies, descriptive norms, and benefits
Behavioral: Expectancies,descriptive norms, benefits, efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies,descriptive norms, benefits, efficacy
Behavioral: Expectancies, descriptive and injunctive norms — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; and correct misperceptions regarding approval of alcohol misuse & sexual risk taking.
  Arms: Expectancies, descriptive and injunctive norms
Behavioral: Expectancies, descr& injun norms, efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies, descr& injun norms, efficacy
Behavioral: Expectancies, desc & injun norms, benefits — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; and increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol.
  Arms: Expectancies, desc & injun norms, benefits
Behavioral: Expectancies,desc & injun norms,benefits,efficacy — Decrease the expectation that alcohol is needed to have good sexual encounter; correct misperceptions of prevalence of alcohol-induced sexual risk behaviors, alcohol use/misuse, and sexual risk behaviors; correct misperceptions regarding approval of alcohol misuse & sexual risk taking; increase perceived benefits to use protective behavioral strategies to reduce the negative consequences of engaging in sexual behaviors under the influence of alcohol; and increase self-efficacy to use protective behavioral strategies (e.g., condom negotiation skills) to reduce unprotected sex.
  Arms: Expectancies,desc & injun norms,benefits,efficacy

SUMMARY:
The overall objective of the proposed research is to reduce the incidence of sexually transmitted infections (STIs) among college students. The investigators propose to accomplish this by using the innovative, engineering-inspired multiphase optimization strategy (MOST) to develop a highly effective, appealing, economical, and readily scalable internet-delivered behavioral intervention targeting the intersection of alcohol use and sexual risk behavior. The rate of STIs on college campuses is alarming: one in four college students is diagnosed with an STI at least once during their college experience. Sexual activity when drinking alcohol is highly prevalent among college students. Alcohol use is known to contribute to the sexual risk behaviors that are most responsible for the transmission of STIs, namely unprotected sex, contact with numerous partners, and "hook-ups" (casual sexual encounters). Few interventions have been developed that explicitly target the intersection of alcohol use and sexual risk behaviors, and none have been optimized. In order to reduce the incidence of STI transmission among this and other high-risk groups, a new approach is needed. MOST is a comprehensive methodological framework that brings the power of engineering principles to bear on optimization of behavioral interventions. MOST enables researchers to experimentally test the individual components in an intervention to determine their effectiveness, indicating which components need to be revised and re-tested. Given the high rates of alcohol use and sex among college students, the college setting provides an ideal opportunity for intervening on alcohol use and sexual risk behaviors. The proposed study will include a diverse population of college students on 4 campuses which will increase the generalizability of the findings. The specific aims are to (1) develop and pilot test an initial set of online intervention components targeting the link between alcohol use and sexual risk behaviors, (2) use the MOST approach to build an optimized preventive intervention, and (3) evaluate the effectiveness of the newly optimized preventive intervention using a fully powered randomized controlled trial (RCT). This work will result in a new, more potent behavioral intervention that will reduce the incidence of STIs among college students in the US, and will lay the groundwork for a new generation of highly effective STI prevention interventions aimed at other subpopulations at risk.

DETAILED DESCRIPTION:
As part of the MOST approach, the investigators will conduct a series of screening experiments to build an optimized intervention. The current study is the first (of two) screening experiments.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled at an American college or University.
* A first year student or first-year transfer student.
* 18 years of age or older.
* Have not gone through previous versions of itMatters before

Exclusion Criteria:

* Not a first year student or transfer student
* Younger than 18 years of age
* Have gone through previous versions of itMatters

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3997 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Descriptive norms about the intersection of alcohol and sex collected via an online questionnaire. | This measure will be assessed immediately following the 3-week intervention
  This scale consists of 6 items and will be created as a weighted scale score. Analyses will report the mean and standard deviation and expected mean values from a regression analysis. The scale will reflect the average perceived prevalence of the alcohol and sex behaviors.
Injunctive norms about the intersection of alcohol and sex collected via an online questionnaire. | This measure will be assessed immediately following the 3-week intervention
  This scale consists of 6 items and will be created as a weighted scale score. Analyses will report the mean and standard deviation and expected mean values from a regression analysis. The scale will reflect the average perceived approval of the alcohol and sex behaviors, ranging from strongly disapprove to strongly approve.
Expectancies about the intersection of alcohol use and sex collected via an online questionnaire. | This measure will be assessed immediately following the 3-week intervention
  This scale consists of 10 items and will be created as a weighted scale score. Analyses will report the mean and standard deviation and expected mean values from a regression analysis. The scale will reflect the average number of drinks expected to experience the 10 different outcomes.
Perceived benefits about using protective behavioral strategies collected via an online questionnaire. | This measure will be assessed immediately following the 3-week intervention
  This scale consists of 11 items and will be created as a weighted scale score. Analyses will report the mean and standard deviation and expected mean values from a regression analysis. The scale will reflect the average likelihood of contracting an STI using the listed behaviors.
Self-efficacy to use protective behavioral strategies collected via an online questionnaire. | This measure will be assessed immediately following the 3-week intervention
  This scale consists of 9 items and will be created as a weighted scale score. Analyses will report the mean and standard deviation and expected mean values from a regression analysis. The scale will reflect the average level of confidence is using protective behavioral strategies to reduce the risk of contracting and STI, ranging from not at all confident to extremely confident.

SECONDARY OUTCOMES:
Binge drinking behavior collected via an online questionnaire | This measure will be assessed 1 month following the completion of the intervention
  This item asks how many times in the past two weeks a male has 5 or more drinks in a 2-hour period (or females 4 or more drinks in a 2-hour period). This variable will be collapsed into 1 or more times versus other and reported as a prevalence of this behavior and used as a dichotomous outcome in regression analyses.
Unprotected sex behavior at most recent sex collected via an online questionnaire | This measure will be assessed 1 month following the completion of the intervention
  This item asks whether or not a condom was used for oral, anal or vaginal sex. This variable will be collapsed into a dichotomous variable with unprotected anal or vaginal sex versus other and reported as a prevalence of this behavior and used as a dichotomous outcome in regression analyses.
Penetrative sex at most recent hookup collected via an online questionnaire | This measure will be assessed 1 month following the completion of the intervention
  This item asks whether or not the most recent hookup included vaginal or anal sex. This variable will be collapsed into a dichotomous variable with penetrative sex versus other and reported as a prevalence of this behavior and used as a dichotomous outcome in regression analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Collins, PhD, Principal Investigator — Penn State University
Locations (4):
- United States (4):
  - Fresno State University, Fresno, California
  - Southern Illinois University, Carbondale, Illinois
  - North Carolina A&T State University, Greensboro, North Carolina
  - North Dakota State University, Fargo, North Dakota

IPD SHARING:
Plan to Share IPD: No